CLINICAL TRIAL: NCT02432885
Title: Myocardial Fibrosis Progression in Duchenne and Becker Muscular Dystrophy - Angiotensin-Converting-Enzyme (ACE) Inhibitor Therapy
Brief Title: Myocardial Fibrosis Progression in Duchenne and Becker Muscular Dystrophy - ACE Inhibitor Therapy Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Collaborators: Federal University of Minas Gerais (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Eduardo Rochitte, Associate Professor of Cardiology, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1095/08
Record Dates: First submitted 2015-03-24; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Myocardial Fibrosis; Muscular Dystrophies
Keywords: cardiac magnetic resonance; myocardial fibrosis; muscular dystrophies
MeSH Terms: conditions — Muscular Dystrophies | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE inhibitor (Experimental): ACE inhibitor (enalapril up to 20mg BID), in patients with preserved EF (LVEF grater than 50%) and with detectable delayed enhancement (myocardial fibrosis) in cardiac magnetic resonance, randomized to therapy or not.
  Interventions: Drug: Enalapril
- Control (No Intervention): Patients with preserved EF (LVEF grater than 50%) and with no detectable delayed enhancement (myocardial fibrosis) in cardiac magnetic resonance

INTERVENTIONS:
Drug: Enalapril — up to 20mg bid
  Arms: ACE inhibitor

SUMMARY:
This trial intends to evaluate myocardial Fibrosis progression in Duchenne and Becker Muscular Dystrophy, as well the influence of ACE inhibitors in fibrosis progression. Additionally, this study aims to determine genetic predictors of cardiac involvement in these dystrophies.

DETAILED DESCRIPTION:
Duchenne and Becker muscular dystrophies (DMD/BMD) are diseases characterized by progressive skeletal muscle degeneration and replacement by fibrofatty tissue. Data on cardiac involvement (defined as myocardial fibrosis), effect of ACE-inhibitors and specific genetic mutations on myocardial involvement detected by cardiac magnetic resonance (CMR) is lacking.

The study will include 76 patients with DMD/BMD. All patients will be referred to two CMRs for assessment of ventricular function and myocardial fibrosis. Patients with myocardial fibrosis and normal left ventricle ejection fraction (LVEF) will be randomized into two groups, each group receiving ACE-inhibitor treatment or no treatment for cardiomyopathy. A genetic profile will be performed in every patient to identify possible mutations related to cardiac involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven Muscular Dystrophy of Duchenne or Becker

Exclusion Criteria:

* Contraindications to cardiovascular magnetic resonance imaging

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quantitative Myocardial Fibrosis by CMR in patients with and without ACE inhibitor therapy | 2 years
  Progression of myocardial fibrosis

SECONDARY OUTCOMES:
Specific genetic mutations as predictors of cardiac involvement | 2 years
  Relation of dystrophin gene site mutations in exons <45 relation and the extent of myocardial fibrosis measured by cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Rochitte, MD, PhD, Principal Investigator — InCor, Heart Institute, University of Sao Paulo Medical School

REFERENCES:
- [Derived] Silva MC, Magalhaes TA, Meira ZM, Rassi CH, Andrade AC, Gutierrez PS, Azevedo CF, Gurgel-Giannetti J, Vainzof M, Zatz M, Kalil-Filho R, Rochitte CE. Myocardial Fibrosis Progression in Duchenne and Becker Muscular Dystrophy: A Randomized Clinical Trial. JAMA Cardiol. 2017 Feb 1;2(2):190-199. doi: 10.1001/jamacardio.2016.4801. PMID 27926769